CLINICAL TRIAL: NCT00492336
Title: Rasagiline in the Treatment of Persistent Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Robert Buchanan, Chief, Maryland Psychiatric Research Center, Outpatient Research Program, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00043807; H-27877 (Other: University of Maryland Baltimore)
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2013-06

CONDITIONS: Schizophrenia
Keywords: Cognitive impairments; Negative symptoms
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rasagiline (Active Comparator): Treatment with Rasagiline
  Interventions: Drug: rasagiline (Pharmacodynamics)
- Inactive pill (Placebo Comparator): Treatment with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rasagiline (Pharmacodynamics) — Rasagiline 1 mg/day for 12 weeks
  Arms: Rasagiline
Drug: Placebo — Placebo 1 tablet each day
  Arms: Inactive pill

SUMMARY:
This is a study of a new medication for the treatment of cognitive impairments (thinking difficulties) and negative symptoms in people with schizophrenia. The new medication is rasagiline. Rasagiline is a drug which has been approved by the Food and Drug Administration for the treatment of Parkinson's disease. It is used to treat cognitive problems.

DETAILED DESCRIPTION:
The study will consist of two phases: a 4-week continued stability phase (lead-in phase) and a 12-week double-blind treatment phase. In the lead-in phase, subjects receiving antipsychotic medication, who manifest moderate to severe and persistent negative symptoms, will remain on their maintenance regimen for at least four weeks. The treatment phase will be a 12-week, parallel groups, double-blind, placebo-controlled trial of adjunctive rasagiline (1 mg/day), a selective MAO-B oxidase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will meet DSM-IV criteria for schizophrenia or schizoaffective disorder.
* Current treatment with one or more second generation antipsychotics, except ziprasidone
* On same second generation antipsychotic(s)for at least 56 days
* On same dose of second generation antipsychotic(s)for at least 30 days
* 22-item SANS: Total score (i.e.all items minus global items and poverty of content of speech)greater than 20 or global Rating of Affective Flattening greater than or equal to 3 or global Rating of alogia greater than or equal to 3
* BPRS: Sum of the four positive symptom items less than or equal to 16 (items 4,11,12,15)
* BPRS: Sum of the four Anxiety/Depression Factor items less than or equal to 14 (items 1,2,5,9)
* Simpson-Angus Scale: Total score less than or equal to 8

Exclusion Criteria:

* DSM-IV Major Depressive Disorder within last 6 months
* Current treatment with ziprasidone
* DSM-IV diagnosis of alcohol or substance dependence within the last 6 months
* DSM-IV criteria for alcohol or substance abuse within the last month
* evidence of illicit substance use, as identified with urine toxicology screen
* History of an organic brain disorder, mental retardation,epilepsy, or a medical condition, whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with the proposed treatment protocol. See those listed below
* Uncontrolled hypertension defined as BP exceeding 145/90 on 3 consecutive readings despite adequate treatment, pheochromocytoma, melanoma, hepatic insufficiency
* Pregnancy or lactation in females
* Pheochromocytoma
* Melanoma
* Hepatic insufficiency

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Buchanan, M.D., Principal Investigator — University of Maryland, College Park
Locations (5):
- United States (5):
  - Baltimore VA Medical Center, Baltimore, Maryland
  - Keypoint Mental health Center, Catonsville, Maryland
  - Maryland Psychiatric REsearch Center, Catonsville, Maryland
  - Mosaic Community Mental health Center, Catonsville, Maryland
  - Keypoint Mental health Center, Dundalk, Maryland

REFERENCES:
- [Derived] Buchanan RW, Weiner E, Kelly DL, Gold JM, Keller WR, Waltz JA, McMahon RP, Gorelick DA. Rasagiline in the Treatment of the Persistent Negative Symptoms of Schizophrenia. Schizophr Bull. 2015 Jul;41(4):900-8. doi: 10.1093/schbul/sbu151. Epub 2014 Nov 2. PMID 25368372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between May 2007-October 2011 from mental health clinics throughout the community.
Pre-assignment Details: Participants were excluded before assignment to treatment groups if they met any of the exclusion criteria, if they became clinically unstable, or they decided that the demands of the study were too great. 84 participants were enrolled into active participation; 57 started study treatment.
Period: Overall Study
Arm/Group | Rasagiline | Inactive Pill
Started | 28 | 29
Completed | 26 | 23
Not Completed | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rasagiline | Inactive Pill | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (12.2) | 45.9 (11.1) | 46.09 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 24 | 22 | 46
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Negative Symptoms
Description: The Scale for the Assessment of Negative Symptoms (SANS) rating scale was used to assess the negative symptoms of schizophrenia. Scores on the subscales are combined (summed) to compute a total score. There are a total of 17 subscales. Each subscale ranges from 0="Not at all" to 5="Severe". Every 4 weeks the summed subscale scores provide a total score for that week (0-85). Higher scores indicate more severe negative symptoms.
Time Frame: Every 4 weeks over a 12 week period
Population: Number of participants available for symptom efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 28
units on a scale
  Week 0 | 32.7 (8.5) | 33.5 (7.8)
  Week 4 | 31.2 (9.4) | 32.3 (8.2)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 31.1 (8.1) | 34.1 (8.6)
  Week 12: number analyzed (Participants) | 26 | 23
  Week 12 | 29.9 (3.9) | 34.3 (8.6)

2. Primary Outcome: Cognitive Testing - Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Score
Description: The RBANS is a brief, individually administered test designed to evaluate neuropsychological status of adults, ages 20-89. The 12 subtests measure attention, language, visuospatial/constructional abilities, and immediate and delayed memory. The raw scores from the subtests are scaled together to create index scores, and these are summed for conversion to a total scale score. Higher score equals a better outcome. The total index score range for the RBANS is 40-160.
Time Frame: Beginning of treatment phase (week 0) and end of treatment phase (week 12)
Population: Subjects completing the cognitive testing at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 23
units on a scale
  Week 0 | 76.8 (12.5) | 74.2 (13.7)
  Week 12 | 78.7 (14.1) | 75.3 (14.5)
  Change | 1.9 (6.9) | 1.1 (7.5)

3. Primary Outcome: Cognitive Testing - N-Back Neurocognitive Task
Description: The N-Back task is a sequential letter working memory task. D-prime was used to measure accuracy on the 0-back, 1-back, and 2-back conditions. D-prime scores range from 0 to 8.6. Higher scores are better. As memory load increases from 0 to 1, from 1 to 2, D-prime scores are expected to be lower.
Time Frame: Beginning of treatment phase (week 0) and end of treatment phase (week 12)
Population: Subjects completing the cognitive testing at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 23
units on a scale
  0-Back: Week 0 | 3.47 (0.74) | 3.52 (0.70)
  0-Back: Week 12 | 3.79 (0.61) | 3.66 (0.71)
  0-Back: Change | 0.32 (0.53) | 0.14 (0.75)
  1-Back: Week 0 | 2.75 (0.73) | 2.63 (0.73)
  1-Back: Week 12 | 2.96 (0.67) | 2.66 (0.91)
  1-Back: Change | 0.20 (0.73) | 0.03 (0.70)
  2-Back: Week 0 | 1.75 (0.72) | 1.56 (0.87)
  2-Back: Week 12 | 1.59 (0.88) | 1.57 (0.86)
  2-Back: Change | -0.16 (0.68) | 0.01 (0.62)

4. Primary Outcome: Cognitive Testing - Probabilistic Learning Task
Description: To assess reward learning, participants used performance feedback to choose the most frequently rewarded item in each of three pairs of stimuli (one pair had reward probabilities: 80% vs 20%; one pair had reward probabilities of 70% vs 30%; one pair had the probabilities of 60% vs 40 %) (PL; Frank et al, 2004). A total of 240 trials were administered so each pair was seen 80 times. Higher scores represent more frequent choices of the optimal stimulus in each pair. The frequencies with which participants repeated an item choice that was rewarded on the previous presentation (win-stay) is also presented as a percentage. Similarly, the lose-shift score is the percentage of times that participants changed their choice for unrewarded items (lose-shift). The win-stay score serves as a measure of the impact of positive feedback on subsequent choices while the lost-shift score serves as a measure of the impact of negative feedback on subsequent choices.
Time Frame: Beginning of treatment phase (week 0) and end of treatment phase (week 12)
Population: Subjects completing the cognitive testing at both time points. Results for lose shifts are calculated for 24 Rasagiline and 22 Placebo participants, due to missing data created by participants who had zero losses (and hence no need to shift) during both the 3rd and 4th blocks of trials.
Measure: Mean (Standard Deviation); unit: percentage of optimal stimuli chosen
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 23
percentage of optimal stimuli chosen
  80 vs 20: Week 0 | 70.8 (23.7) | 69.1 (25.1)
  80 vs 20: Week 12 | 70.4 (24.5) | 68.5 (25.8)
  80 vs 20: Change | -0.4 (33.8) | -0.7 (36.8)
  70 vs 30: Week 0 | 69.7 (22.3) | 66.1 (19.8)
  70 vs 30: Week 12 | 64.4 (23.4) | 65.9 (18.8)
  70 vs 30: Change | -5.3 (27.4) | -0.2 (25.6)
  60 vs 40: Week 0 | 53.9 (26.9) | 57.9 (24.9)
  60 vs 40: Week 12 | 58.7 (23.8) | 58.6 (18.2)
  60 vs 40: Change | 4.7 (43.0) | 0.7 (29.8)
  Lose Shifts: Week 0: number analyzed (Participants) | 24 | 22
  Lose Shifts: Week 0 | 48.6 (16.4) | 56.5 (12.9)
  Lose Shifts: Week 12: number analyzed (Participants) | 24 | 22
  Lose Shifts: Week 12 | 50.1 (16.9) | 54.8 (12.0)
  Lose Shifts: Change: number analyzed (Participants) | 24 | 22
  Lose Shifts: Change | 2.9 (17.2) | -1.2 (14.9)
  Win Stays: Week 0 | 64.6 (19.5) | 62.2 (18.7)
  Win Stays: Week 12 | 62.9 (20.5) | 64.4 (15.2)
  Win Stays: Change | -1.7 (27.7) | 2.3 (21.9)

5. Primary Outcome: Cognitive Testing - Delayed Discounting
Description: The monetary choice questionnaire for hypothetical monetary rewards was used to assess delayed discounting (Kirby et al, 1999). The measure includes 27 items in which participants choose between a smaller, immediate reward (SIR) and a larger, delayed reward (LDR). There are three LDR sizes: small ($25-35), medium ($50-60) and large ($75-85). By examining the pattern of choices that participants make across the set of 27 items it is possible to calculate their delay discounting rate, termed K. The discount rate determines the steepness of the reduction in the present value of a reward with increases in the delay to the possible receipt of that reward. Thus, higher values in K represent greater discounting of the value of future rewards. With this measure K values can range between a low of 0.00016 to a high of 0.25. Higher K values have been linked to measures of impulsivity. Shown in the table are the K values observed when the future rewards were small, medium, or large.
Time Frame: Beginning of treatment phase (week 0) and end of treatment phase (week 12)
Population: Subjects completing the cognitive testing at both time points.
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 23
units on a scale
  Large Reward: Week 0 | 0.004 [0.001 to 0.010] | 0.018 [0.007 to 0.046]
  Large Reward: Week 12 | 0.010 [0.004 to 0.025] | 0.010 [0.004 to 0.023]
  Medium Reward: Week 0 | 0.003 [0.001 to 0.007] | 0.024 [0.009 to 0.061]
  Medium Reward: Week 12 | 0.008 [0.003 to 0.019] | 0.011 [0.004 to 0.027]
  Small Reward: Week 0 | 0.009 [0.003 to 0.022] | 0.023 [0.011 to 0.048]
  Small Reward: Week 12 | 0.016 [0.006 to 0.043] | 0.014 [0.005 to 0.034]

6. Secondary Outcome: Extrapyramidal Symptoms
Description: The Simpson Angus Scale (SAS; Simpson and Angus, 1970) was used to assess extrapyramidal symptoms (EPS). The assessment consists of 11 items, each rating the severity of potential symptoms of movement disorders. Total scores are calculated by summing the scores of each of the 11 items for a potential total score of 0-44, with higher scores indicating more severe EPS.
Time Frame: Baseline (Week 0) and End of Study (Week 12)
Population: SAS scores were collected at baseline on 28 Rasagiline and 29 Placebo patients. End of study scores were collected on 27 Rasagiline and 27 Placebo patients, including 5 patients who withdrew before Week 12 (1 Rasagiline patient at Week 4, 1 Placebo participant each at Weeks 3 and 6, and two Placebo participants at Week 8).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 28 | 29
units on a scale
  Week 0 | 1.82 (2.30) | 1.93 (2.07)
  Week 12: number analyzed (Participants) | 27 | 27
  Week 12 | 0.96 (1.34) | 1.89 (2.71)
  Change | -0.85 (1.94) | -0.04 (2.24)

7. Secondary Outcome: Number of Participants With Akathisia
Description: The Barnes Akathisia Scale (BAS; Barnes, 1989) was used to assess akathisia, a type of extrapyramidal symptom. The global clinical assessment of akathisia score is rated on a scale from 0=Absent to 5=Severe Akathisia.
Time Frame: Baseline and every two weeks throughout the double-blind phase of the study, for up to 12 weeks.
Population: Barnes Akathisia Scales at baseline and end of study were collected for 26 participants each in the rasagiline and placebo groups. End of study ratings were collected at week 12, except for 4 placebo participants (1 participant each at weeks 3 and 6, and two at week 8).
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 26
Participants
  Score 0=Absent : Baseline | 20 | 21
  Score 0=Absent : End of Study | 20 | 21
  Score 1=Questionable : Baseline | 3 | 5
  Score 1=Questionable : End of Study | 2 | 5
  Score 2=Mild Akathisia : Baseline | 2 | 0
  Score 2=Mild Akathisia : End of Study | 3 | 0
  Score 3=Moderate Akathisia : Baseline | 1 | 0
  Score 3=Moderate Akathisia : End of Study | 1 | 0

8. Secondary Outcome: Change in Persistent Positive Symptoms
Description: The Brief Psychiatric Rating Scale (BPRS) positive symptom item total score was used to assess positive symptom change. The BPRS positive symptom items are: conceptual disorganization, hallucinatory behavior, unusual thought content, and suspiciousness. The total score is calculated by adding the scores for each item. Each scale ranges from "1=Not Present" to "7=Very Severe". The minimum score is 4 and the maximum score is 28. A higher score indicates a more severe positive symptom rating.
Time Frame: Every 4 weeks for 12 weeks.
Population: Number of participants available for symptom efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 28
units on a scale
  Week 0 | 8.8 (3.2) | 9.1 (4.0)
  Week 4 | 9.2 (3.7) | 9.1 (3.9)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 9.2 (3.5) | 9.8 (4.2)
  Week 12: number analyzed (Participants) | 26 | 23
  Week 12 | 8.3 (3.3) | 8.9 (3.7)

9. Secondary Outcome: Depressive Symptoms
Description: The Calgary Depression Scale (CDS; Addington et al, 1997) total score was used to assess depressive symptoms over the course of the study. Total scores were calculated by summing the scores of each of the 9 items. Total scores can range from 0-27, with higher scores indicating more severe depressive symptoms.
Time Frame: Every 4 weeks for 12 weeks.
Population: Number of participants available for symptom efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 28
units on a scale
  Week 0 | 2.29 (2.08) | 2.02 (2.37)
  Week 4 | 2.19 (2.08) | 1.96 (2.30)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 2.31 (1.93) | 1.52 (1.94)
  Week 12: number analyzed (Participants) | 26 | 23
  Week 12 | 2.58 (2.63) | 1.52 (2.25)

10. Secondary Outcome: Global Change in Illness Severity
Description: The Clinical Global Impression (CGI) severity of illness item was used to assess global changes. Scores on this item range from 1="Normal, not at all ill" to 7="Among the most extremely ill".
Time Frame: Every 4 weeks for 12 weeks.
Population: Number of participants available for symptom efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 26 | 28
units on a scale
  Week 0 | 4.05 (0.42) | 4.31 (0.49)
  Week 4 | 4.08 (0.39) | 4.32 (0.48)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 1.00 (0.4) | 4.36 (0.49)
  Week 12: number analyzed (Participants) | 26 | 22
  Week 12 | 1.08 (0.48) | 4.27 (0.46)

11. Secondary Outcome: Number of Participants Exhibiting Side Effects
Description: The Side Effect Checklist (SEC) was used to assess side effects. The SEC is comprised of 22 common side effects, which are rated on a 1 (none)-4 (severe) scale. Side effects are determined to be clinically significant if there is a two or more point increase in severity from baseline, or any side effect that receives a severity rating of "4" (severe) at any point in the treatment phase of the study.
Time Frame: Every week for 12 weeks
Population: One placebo patient for whom a baseline side effects checklist was excluded from these analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Rasagiline | Inactive Pill
Number analyzed (Participants) | 28 | 28
Participants
  Abdominal Pain | 5 | 7
  Anorexia | 7 | 10
  Bruising Easily | 4 | 1
  Constipation | 12 | 9
  Diarrhea | 9 | 6
  Dizziness | 5 | 7
  Dry Mouth | 7 | 11
  Enuresis | 4 | 3
  Fever | 2 | 5
  Headache | 7 | 8
  Hypersalivation | 4 | 7
  Insomnia | 2 | 7
  Malaise | 8 | 14
  Mucosal Ulceration | 1 | 1
  Nausea | 6 | 2
  Rash | 3 | 5
  Restlessness | 4 | 7
  Sedation | 8 | 8
  Sore Throat | 3 | 5
  Stiffness | 7 | 5
  Tremor | 3 | 11
  Urticaria | 3 | 5
  Vomiting | 4 | 4
  Weight Loss | 10 | 12

ADVERSE EVENTS:
Time Frame: During the 12-week Treatment Phase of the study.
Arm/Group | Rasagiline | Inactive Pill
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/29
Other Adverse Events (participants affected / at risk) | 1/28 | 3/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rasagiline (N=28) | Inactive Pill (N=29)
Hospitalization (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rasagiline (N=28) | Inactive Pill (N=29)
suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
increased urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
conceptual disorganization (Psychiatric disorders) | 0 (0) | 1 (1)
tooth problems (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No